CLINICAL TRIAL: NCT04164875
Title: Fever During Labour
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Kim Wildgaard, MD, MD, ph.d.,Clinical Professor, Herlev Hospital
Other Study IDs: 2019 Fever during Labour
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Fever; Due to Heat; Infection
Keywords: fever; epidural; birth; labour
MeSH Terms: conditions — Fever; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Temperature measurement — The 'intervention' is repeated rectal temperature measurements
  Other Names: Fever

SUMMARY:
Pilot study to assess fever during labour.

DETAILED DESCRIPTION:
200 parturients will be monitored for fever during labour using rectal thermometer.

Repeated measurements 1/hr during the first 6 hours will allow us to find patients developing fever.

Fever = rectal temp >38 Celsius twice within 60 min or 39 degrees Celsius measured once .

After birth, blood samples are assessed for infection. Use of Antibiotics and other medication is Recorded. Subgroup analyses based on suspected causes of fever during birth.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, planned vaginal birth, able to give consent

Exclusion Criteria:

* do not speak Danish or English, unable to cooperate to rectal temperature measurements,

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Fever | during labour
  Fever = rectal temp >38 Celsius twice within 60 minutes or 39 degrees Celsius measured once

SECONDARY OUTCOMES:
CRP | 24 hours
  infection marker
Leucocytosis | 24 hours
  infection marker
bacterial growth blood | 1 week
  infection marker
bacterial growth placenta blood | 1 week
  infection marker

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wildgaard, MD phd, Study Chair — Herlev Hospital, Afdeling for Bedøvelse og Operation; Lærke Vinberg Rasmussen, Principal Investigator — Herlev Hospital, Dept. of Obstetriscs
Locations (1):
- Department of Anaesthesiology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No